CLINICAL TRIAL: NCT03872297
Title: Effect of a Fish Collagen Peptide Food Supplement on the Weight and Body Composition of Healthy Volunteers in Overweight
Brief Title: Fish Collagen Peptide Food Supplement on Weight and Body Composition
Acronym: NATICOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, MD in nutrion and endocrinology, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-A02490-55
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Weight Management; Food Complement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo supplement (Placebo Comparator): Consumption of a non active food complement during 3 months.
  Interventions: Dietary Supplement: Placebo supplement
- Naticol supplement (Active Comparator): Consumption of the active food complement during 3 months containing Naticol.
  Interventions: Dietary Supplement: Naticol supplement

INTERVENTIONS:
Dietary Supplement: Placebo supplement — Consumption of a non active food complement during 3 months.
  Tests performed :
  * 2 blood tests :
  * 2 body composition analysis via Dual-energy X-ray absorptiometry (DXA)
  * 2 stool collections The first one of these analysis was performed at the beginning, second at the end of the study.
  Arms: Placebo supplement
Dietary Supplement: Naticol supplement — Consumption of the active food complement during 3 months containing Naticol.
  Tests performed :
  * 2 blood tests :
  * 2 body composition analysis via Dual-energy X-ray absorptiometry (DXA)
  * 2 stool collections The first one of these analysis was performed at the beginning, second at the end of the study.
  Arms: Naticol supplement

SUMMARY:
Fish collagen hydrolysates or peptides orally administered have been investigated in recent clinical trials in human health. These peptides have been evaluated in various biological and medical fields including skin aging, osteoarticular apparatus, muscle and more recently in energy metabolism in both animals and humans.

However, very few studies investigated the effect of fish collagen peptides on weight, body composition or glycemic response. Recently, it has been shown that the consumption of fish collagen peptides (Naticol®) limits weight gain and increase in fat mass in a mouse model made obese by a hyperlipidic diet. Since these results have never been observed in humans, this pilot study proposes to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Men in overweight (BMI between 25kg/m² and 30kg/m²)
* Aged from 18 and 60 years
* Having signed the informed consent form;
* Susceptible to follow the constraints generated by the study;

Exclusion Criteria:

* Subject treated for type 1 or 2 diabetes, or for any other metabolic disorder (severe dyslipidemia: TG> 3 g / L and total cholesterol> 2.5 g / L);
* Subject with untreated and uncorrected high blood pressure;
* Subject with untreated or uncorrected dysthyroidism by drug therapy;
* Subject with a serious general illness that may prevent his or her ability to complete the trial or that could bias the results of the study;
* Subject consuming antibiotic treatment in the month prior to inclusion;
* Subject treated with steroidal anti-inflammatory drugs, anabolic steroids, anticoagulants or corticosteroids;
* Subject knowing allergy to fish or fish collagen;
* Subject taking any dietary supplement or drug that may interact with the results of the study or that could alter the bioavailability of the product under study;
* Subject following or having followed a low-calorie diet (energy intake <1500 kcal / day) in the 3 months preceding inclusion and / or likely to undertake this diet during the test;
* Subject having lost more than 5% of his initial weight during the last 3 months;
* Subject following a special diet: eg. vegetarian, macrobiotic diet, high protein diet;
* Subject with diagnosed eating disorders (anorexia, bulimia);
* Subject with gastrointestinal malabsorption such as celiac disease, Crohn's disease or lactose intolerance;
* Subject having undergone bariatric surgery;
* Subject with excessive alcohol consumption at more than 3 drinks a day ;
* Subject planning to modify his tobacco consumption (eg weaning) or his level of physical activity (significant increase) before the end of the intervention period;
* Subject having an aversion to the grapefruit aroma;
* Subject unable to understand or adhere to the protocol;
* Subject participating in another clinical study or exclusion period from another study;

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To avoid action of femal hormone, this pilot study is based on male population
Enrollment: 40 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Weight of participants | 0 and 3 months
  Weight is expressed in kilograms

SECONDARY OUTCOMES:
Body composition par DXA analysis | 0 and 3 months
  Fat mass is expressed in kg and percent, muscle mass in kg and percent.
Waist circumference | 0 and 3 months
  Data are expressed in centimeters
Lipid profile in plasma | 0 and 3 months
  Total cholesterol, HDL cholesterol, LDL cholesterol, and Triglycerides. Data are expressed in g/L and in mmol/L
Glycemia level in plasma | 0 and 3 months
  Data are expressed in g/L and mmo/L
Insulin level in plasma | 0 and 3 months
  Data are expressed in μU/ml
HOMA index | 0 and 3 months
  This index indicates the insulin resistance and was calculated as follow : HOMA [(glycémie mmol/l X insulinémie μU/ml) à jeun / 22,5]
Physical activity intensity | 0 and 3 months
  Score obtained via Ricci and Gagnon questionnaire. The questionnaire contains 9 questions ; score could be between 9 and 45 points.
  * under 18 points : inactive behavior
  * between 19 and 35 points : active behavior
  * over 35 points : very active behavior
Pro-inflammatory cytokines concentration | 0 and 3 months
  Assay for TNFalpha, IL-1beta and IL-6 in plasma
Microbiota analysis | 0 and 3 months
  Rate comparison of different bacteria families
Height | 0
  centimeters
Body mass index | 0 and 3 months
  kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No